CLINICAL TRIAL: NCT05636735
Title: Self-confidence in Midwife Students
Acronym: ESF-conf
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_RIPH_015_ESF-conf
Record Dates: First submitted 2022-11-22; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Midwife Students
Keywords: midwife students; self-confidence; stress
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- midwife students group: midwife students in France
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — evaluation of self -confidence

SUMMARY:
Self-confidence is essential during the training of students but in professional practice. Therefore, the training of students must allow its acquisition.

However, the university environment is particularly stressful for students. This stress can lead to depression. Perceived stress refers to the feeling of inability to pass an exam even if the person has the abilities to do so.

DETAILED DESCRIPTION:
aim of the study is to describe the level of self-confidence of midwife students.

ELIGIBILITY:
Inclusion Criteria:

* midwife students
* with or without repeating a grade
* in France
* agreeing to participate in the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: midwife students
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-01-17 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
self-confidence | day 0
  self-confidence evaluated using 13 questions about professional abilities (to be able to diagnostic, for example). Each question is coded on a 4-point scale (totally disagree / tend to disagree / tend to agree / totally agree) for a score ranging from 13

CONTACTS AND LOCATIONS:
Locations (1):
- Ufr Medecine Urca, Reims, France

IPD SHARING:
Plan to Share IPD: No